CLINICAL TRIAL: NCT06655974
Title: Protocol for Evaluating the Effectiveness of a Clinical Decision Support System With Prediction Modeling to Identify Patients With Health-related Social Needs in the Emergency Department
Brief Title: Predictive Modeling for Social Needs in Emergency Department Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Joshua R. Vest, PhD, Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011558232
Record Dates: First submitted 2024-08-23; First posted 2024-10-24 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Emergency Service, Hospital; Social Determinants of Health
Keywords: informatics
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: The intervention will be at the ED level using a pre-post design with a matched comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision support intervention group (Experimental): Adult ED patients seeking care the ED site with the health-related social needs decision support system live.
  Interventions: Other: Health-related social needs decision support system
- Comparison group (No Intervention): Adult ED patients created using statistical matching from ED sites in the same metropolitan area.

INTERVENTIONS:
Other: Health-related social needs decision support system — The clinical decision support intervention will present emergency department clinicians at an Indianapolis, IN ED with a likelihood score for an adult patient screening positive for the following health-related social needs (HRSNs): housing instability, food insecurity, transportation barriers, financial strain, and history of legal involvement. For each HRSN, the likelihood of screening positive is reported as "high", "medium", or "low". These categorizations are the product of logistic regression models. The clinical decision support intervention will be delivered through an existing FHIR (Fast Healthcare Interoperability Resources) standards-based clinical decision support platform.
  Arms: Decision support intervention group

SUMMARY:
The overall objective of this study is to support emergency department management of patients' health-related social needs. This study will measure the impact of a decision support system that informs clinicians about which patients are likely to screen positive for a health-related social need. The system uses statistical models to create a health-related social need risk score for each patient. The main questions, the study aims to answer are:

* Does providing emergency department clinicians with risk scores on health-related social needs increase screening and referral activities?
* Does providing emergency department clinicians with risk scores on health-related social needs change patients' use of healthcare services?

The decision support system with health-related social needs risk scores will be introduced for all adult patients at one emergency department. Screening rates, referrals, and subsequent healthcare encounters will be compared with emergency departments that did not have access to the decision support system.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years old)
* Seeking care at Indianapolis, Indiana area emergency departments (EDs).

Exclusion Criteria:

* Children
* Encounters by patients that present with a critical illness/injury (e.g. severe trauma patients or those with Emergency Severity Index (ESI) classification level 1)
* Encounters by patients who have been transferred from another inpatient facility
* Patients that die during the ED encounter
* Encounters among patients who were ultimately admitted during their ED visits from our analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48000 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent of emergency department encounters screened for health-related social needs (HRSNs) | At time of emergency department encounter (or within 24 hours)
  The numerator will be an emergency department encounter with any indication of HRSN screening using any tool or questionnaire, regardless of patient completion or results. The denominator will be all eligible ED encounters.
Percent of emergency department encounters that were referred for health-related social needs (HRSNs) services | At time of emergency department encounter (or within 24 hours)
  The numerator will be emergency department encounters with a referral to social worker, case management, community health workers, or related services within 24 hours of the ED encounter. The denominator will be all eligible ED encounters

SECONDARY OUTCOMES:
Percent of encounters with an emergency department revisit measured at 3 days | within 3 days of emergency department encounter
  The numerator will be an emergency department encounter at any facility included in the Indiana for Network Care database within 3 days of an ED encounter at an intervention or comparator site. ED revisits may serve as the index visit for subsequent revisits. The denominator will be all eligible ED encounters. Encounters resulting in an inpatient admission will be excluded from the numerator and denominator.
Percent of encounters with an emergency department revisit measured at 7 days | within 7 days of emergency department encounter
  The numerator will be an emergency department encounter at any facility included in the Indiana for Network Care database within 7 days of an ED encounter at an intervention or comparator site. ED revisits may serve as the index visit for subsequent revisits. The denominator will be all eligible ED encounters. Encounters resulting in an inpatient admission will be excluded from the numerator and denominator.
Percent of encounters with an emergency department revisit measured at 30 days | within 30 days of emergency department encounter
  The numerator will be an emergency department encounter at any facility included in the Indiana for Network Care database within 30 days of an ED encounter at an intervention or comparator site. ED revisits may serve as the index visit for subsequent revisits. The denominator will be all eligible ED encounters. Encounters resulting in an inpatient admission will be excluded from the numerator and denominator
Percent of emergency department encounters with primary care visit within 7 days of an ED encounter | within 7 days of emergency department visit
  The numerator will include all emergency department encounters with a completed family medicine, internal medicine, OBGYN, or geriatrician visit64 within 7 days of the ED visit. The denominator will be all eligible ED encounters. Encounters resulting in an inpatient admission will be excluded from the numerator and denominator.

OTHER OUTCOMES:
Percent of emergency department encounters where the health-related social needs (HRSN) decision support system intervention was accessed. | At time of emergency department encounter (or within 24 hours)
  The numerator will include encounters with access of the social needs section (containing the risk prediction scores) of the decision support system intervention during the study visit (defined as within 24 hours). Access will be defined as record of the end user visiting the HRSN page in the system user logs. The denominator will be all eligible ED encounters. Limited to the intervention site only.
Percent of emergency department encounters where the clinical decision support platform was accessed | At time of emergency department encounter(or within 24 hours)
  The numerator will include encounters with access of clinical decision support platform during the study visit (defined as within 24 hours). Access will be defined as record of the end user visiting initiating a request to the decision support application from the EHR. Any portion of the decision support platform (not just the health-related social needs section) is included. The denominator will be all eligible ED encounters (see Inclusion criteria, above). Limited to the intervention site only

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Vest, PhD,MPH, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
All data produced during the project will be preserved, but raw and derived data (at the patient-level) will not be posted publicly because of our use of secondary data from privately held electronic health record and health information exchange systems. Due to the data use restrictions put in place by consortium agreements among the health system partners that contribute EHR data to the Indiana Network for Patient Care, patient-level data cannot be shared or disseminated outside this project. However, de-identified derived data (at the patient-level) used in this study may be shared with investigators whose formal request is approved by the data owners. Requests can be sent to askRDS@regenstrief.org. Access to these data requires investigator support for use and a signed data access agreement between the Regenstrief Institute and the investigator's institution.

REFERENCES:
- [Background] Mazurenko O, Hirsh AT, Harle CA, McNamee C, Vest JR. Acceptance of Automated Social Risk Scoring in the Emergency Department: Clinician, Staff, and Patient Perspectives. West J Emerg Med. 2024 Jul;25(4):614-623. doi: 10.5811/westjem.18577. PMID 39028248
- [Derived] Mazurenko O, Harle CA, Blackburn J, Menachemi N, Hirsh A, Grannis S, Boustani M, Musey PI Jr, Schleyer TK, Sanner LM, Vest JR. Effectiveness of a clinical decision support system with prediction modeling to identify patients with health-related social needs in the emergency department: Study protocol. PLoS One. 2025 May 12;20(5):e0323094. doi: 10.1371/journal.pone.0323094. eCollection 2025. PMID 40354398